CLINICAL TRIAL: NCT02148835
Title: Influence of Dietary Omega-3 Fatty Acids in Various triOMEG Sausages on the HS-Omega-3 Index in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemens von Schacky (Other)
Collaborators: Südbayerische Fleischwaren GmbH (Unknown)
Responsible Party: Sponsor-Investigator, Clemens von Schacky, Sponsor-Investigator, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 543-13
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
Keywords: Omega-3 Index; Bioavailability; Eicosapentaenoic acid; Docosahexaenoic acid; Fortified food

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triomeg (Active Comparator): Sausage: Triomeg
  Interventions: Other: Sausage: Triomeg
- Control sausage (Placebo Comparator): Sausage: Control
  Interventions: Other: Sausage: Control

INTERVENTIONS:
Other: Sausage: Triomeg — Commercial sausages enriched with 330 - 510 mg EPA+DHA / 100 g Approximate average composition of active product per 80 g Sausage (Triomeg): 250 mg EPA+DHA as ethyl-ester Energy content 500 kJ (120 kcal), protein 12 g, Carbohydrates 0.8 g, total fat 9 g, of which 2.8 g saturated fatty acids, 4.5 g monounsaturates, 1.4 g polyunsaturates. sodium 0.66 g.
  Arms: Triomeg
Other: Sausage: Control — Control sausage: as active, but no EPA+DHA ethyl-ester.
  Arms: Control sausage

SUMMARY:
New approaches to increase eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in our diet are needed, but any new approach needs to demonstrate the bioavailability of EPA+DHA, and its safety and palatability. The HS-Omega-3 Index is a prime parameter to demonstrate bioavailability in the long-term. Study hypothesis is that increased intake of EPA+DHA will increase the HS-Omega-3 Index. Study aim is to investigate how supplementing various sausages with omega-3 fatty acids influences the HS-Omega-3 Index in healthy volunteers, as compared to unsupplemented matching sausages. Safety and palatability of the sausages are also to be assessed.

DETAILED DESCRIPTION:
Randomized, placebo-controlled, mono-center comparison of two matching groups of sausages (active vs. control). The study will be conducted according to Good Clinical Practice. Randomization will be computer-generated by the sponsor. Sealed envelopes will be provided to the Investigator bearing individual randomization numbers, containing individual randomization results. Thus, in case of need, one sealed envelope can be opened to learn the randomization result of one patient without overall unblinding.

Study participants will be requested to ingest approx. 80 g / day of the experimental sausages during the day at a time of their convenience. Study participants will be provided with the investigational product free of charge. If necessary, the investigational product will be shipped to study participants. Study participants will receive the exact amount of sausages to complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing to eat 80 g of the sausage to be investigated per day.
2. Age: 20 - 60 years
3. Low HS-Omega-3 Index (<5%)
4. Subjects must have adequate fluency in German or English to complete baseline and follow-up interviews.
5. Stable intake of food containing EPA+DHA before and during study
6. Subjects must be able and willing to give written informed consent, and to comply with study procedures.

Exclusion Criteria:

1. Subjects for whom the intake of omega-3 fatty acids is mandatory according to recent treatment guidelines or who take omega-3 fatty acids supplements on a regular basis.
2. Subjects consuming >2 portions of fatty fish / week
3. Subjects with serious bleeding disorder. Use of platelet inhibitors or conventional anticoagulation with a target INR of 2.0 - 3.0 is not an exclusion criterion.
4. Subjects with any acute and life-threatening condition, such as collapse and shock, acute myocardial infarction (last three months), stroke, embolism.
5. Subjects with significant medical co-morbidity, seriously limiting life expectancy or insulin-treated diabetes mellitus or a BMI>30
6. Allergy/intolerance or history of hypersensitivity to components of study intervention.
7. Pregnant subjects and breastfeeding subjects. In addition, women of childbearing potential who will not practice a medically accepted method of contraception will be excluded.
8. Subjects who, in the investigator's judgement, will not likely be able to comply with the study protocol or with known drug- or alcohol abuse/dependence in the past 2 years.
9. Use of any investigational agents within 30 days prior to t0

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anton Köhler, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Dept. of Preventive Cardiology, Ludwig Maximilians-University Munich, Munich, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triomeg | Control Sausage
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Triomeg | Control Sausage | Total
Number analyzed (Participants) | 22 | 22 | 44
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (8.0) | 25.6 (4.1) | 26.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: HS-Omega-3 Index at Baseline and End of Study
Description: The HS-Omega-3 Index is the percentage of EPA+DHA in erythrocytes, as assessed with a highly standardized analytical procedure. Since the HS-Omega-3 Index correlates with tissue EPA+DHA, it represents an individual's status in EPA+DHA.
Time Frame: baseline and 8 weeks
Population: As recruited.
Measure: Mean (Standard Deviation); unit: HS-Omega-3 Index
Arm/Group | Triomeg | Control Sausage
Number analyzed (Participants) | 22 | 22
HS-Omega-3 Index
  baseline | 4.18 (0.54) | 4.32 (0.35)
  8 weeks | 5.72 (0.66) | 4.50 (0.51)

2. Secondary Outcome: Safety and Palatability of the Study Sausage
Description: Serious adverse events (SAE) not necessarily ending study participation are:
  * hospitalizations and surgical procedures
  * life-threatening events and accidents
  * Events leading to permanent damage to study participants,
  Moreover, all other medical events will be recorded. All events qualifying as AE or SAE, according to Good Clinical Practice, will be recorded and reported to the ethic´s committee.
Time Frame: 10 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 Weeks
Arm/Group | Triomeg | Control Sausage
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 4/22 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triomeg (N=22) | Control Sausage (N=22)
Minor adverse events (Gastrointestinal disorders) | 0 (0) | 1 (1) — One participant had mild GI symptoms not related to the investigational product, considered not related to the investigational product.
Minor adverse event (Gastrointestinal disorders) | 0 (0) | 1 (1) — One participant had a viral infection with fever, diarrhea and emesis, considered not related to the investigational product.
Minor adverse event (Infections and infestations) | 1 (1) | 0 (0) — One participant had influenza, considered not related to the investigational product.
Minor adverse event (Infections and infestations) | 3 (3) | 0 (0) — Three participants had mild symptoms of a cold, considered not related to the investigational product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No